CLINICAL TRIAL: NCT03363425
Title: Effect of Perioperative Intravenous Infusion of Dexmedetomidine vs. Lidocaine on Postoperative Pain, Analgesic Consumption, Bowel Function and Recovery After Abdominal Gynaecological Surgery: a Randomised Double Blind Study
Brief Title: Effect of Perioperative iv Dexmedetomidine vs. Lidocaine on Postoperative Pain, Analgesic Consumption and Recovery After Abdominal Gynaecological Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Staikou Chryssoula, Assistant Professor of Anaesthesiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EE-2/04/31-01-2017
Record Dates: First submitted 2017-11-23; First posted 2017-12-06 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Hysterectomy; Myomectomy
Keywords: Dexmedetomidine; Lidocaine; Postoperative Pain; Analgesic Consumption; Recovery; Abdominal Gynaecological Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine Iv
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Normal Saline 0,9% (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine Iv — Lidocaine Iv
  Arms: Lidocaine
Drug: Dexmedetomidine — dexmedetomidine iv
  Arms: Dexmedetomidine
Drug: Normal saline — placebo
  Arms: Normal Saline 0,9%

SUMMARY:
Postoperative pain continues to be inadequately managed and is the most common reason for the delay in discharge and unplanned hospital admission after surgery. Opioids remain the mainstay for postoperative analgesia. However, there is a continuous search for adjuvant therapies to reduce the doses of opioids and their related adverse effects, and extend the use of non-opioid analgesia for acute pain after abdominal surgery, thereby improving patient recovery. Currently there are no clinical trials that investigate the effect of intravenous lidocaine vs dexmedetomidine on postoperative pain, analgesic consumption and bowel function of patients undergoing abdominal gynaecological surgery. Purpose of this prospective double blind randomised clinical trial is the investigation of the effect of perioperative intravenous infusion of lidocaine vs dexmedetomidine vs placebo (Normal Saline 0,9%) on analgesic parameters and functional recovery of patients undergoing abdominal gynaecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* women
* ASA I-II
* 30-70 years
* abdominal gynaecological surgery

Exclusion Criteria:

* patient's refusal
* contraindication to the use of local anesthetics
* body mass index >30 kg/m2
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* pregnant women
* significant renal or hepatic impairment
* insulin-dependent diabetes mellitus
* central nervous system disease or psychiatric diseases
* chronic use of opioids, steroids, clonidine (or other a2 agonist)
* use of drugs acting on the central nervous system or analgesics during the previous 2 weeks
* drug/alcohol abuse
* inability to comprehend the following pain assessment scale

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
analgesic consumption 24 hours postop | 24 hours postoperatively
  morphine consumption from PCA

SECONDARY OUTCOMES:
postoperative pain | 0 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)
postoperative pain | 2 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)
postoperative pain | 4 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)
postoperative pain | 8 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)
postoperative pain | 24 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)
postoperative pain | 48 hours postoperatively
  Numeric Pain Rating Scale- NPRS scale (0:no pain 10:worst pain ever)

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieio University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rekatsina M, Theodosopoulou P, Staikou C. Perioperative Dexmedetomidine or Lidocaine Infusion for the Prevention of Chronic Postoperative and Neuropathic Pain After Gynecological Surgery: A Randomized, Placebo-Controlled, Double-Blind Study. Pain Ther. 2022 Jun;11(2):529-543. doi: 10.1007/s40122-022-00361-5. Epub 2022 Feb 15. PMID 35167059
- [Derived] Rekatsina M, Theodosopoulou P, Staikou C. Effects of Intravenous Dexmedetomidine Versus Lidocaine on Postoperative Pain, Analgesic Consumption and Functional Recovery After Abdominal Gynecological Surgery: A Randomized Placebo-controlled Double Blind Study. Pain Physician. 2021 Nov;24(7):E997-E1006. PMID 34704710